## **Medtronic**

161 Cheshire Lane Suite 100 Plymouth, MN 55441 USA www.medtronic.com

Official Title: A Post-market Feasibility Study Evaluating Location Accuracy Using the superDimension™ Navigation System Version 7.2 With Fluoroscopic Navigation Technology in Subjects Undergoing Lung Lesion Biopsy

ClinicalTrials.gov ID: NCT03585959

Date of Document: 05Dec2019

## **Note to File Fluoroscopic Navigation Study**

**GBET-091** 

v2

Page 1 of 2



## **Note to File**

| Study name: | MDT18004ILSFNV<br>(Fluoroscopic Navigation<br>Clinical Study) | Investigation Site Name/ Number (if applicable): | N/A |
|---|---|---|---|
| Subject: | Fluoroscopic Navigation Clinical Study Inclusion/Exclusion Criteria CIP Typos | | |

| Prepared by | Katie Bayliss |
|---------------------|------------------------------------------------|
| Date of preparation | 20 Nov 2019 |
| Document | Fluoroscopic Navigation CIP_Final_v1.0_09Apr18 |

This Note to File is to document typos in the inclusion and exclusion criteria of the Clinical Investigation Plan (CIP) for the Fluoroscopic Navigation Clinical Study.

On 18Sep19 the ILS Medical Writer identified a typo in the CIP for the Fluoroscopic Navigation Clinical Study regarding the Exclusion Criteria 1. The word "not" was included in error:

Central lesions that are **not** visible endobronchially or could be reached by a flexible bronchoscope or endobronchial ultrasound (EBUS) without utilization of ENB

Exclusion Criteria 1 should have stated: ee K. Baylin 5 Dec 2019

Central lesions that are <del>not</del> visible endobronchially or could be reached by a flexible bronchoscope or endobronchial ultrasound (EBUS) without utilization of ENB



On 29Oct19, a site Principal Investigator noticed that Inclusion Criteria 1 inaccurately states the targeted lesion size for protentional subjects:

Subjects presents with lung lesion(s) greater than 10 mm in diameter amendable to evaluation by the ENB at the time of the evaluation

Inclusion Criteria 1 should have stated:

## **Note to File Fluoroscopic Navigation Study**



v2

Page 2 of 2



Subjects presents with lung lesion(s) greater than *or equal to* 10 mm in diameter amendable to evaluation by the ENB at the time of the evaluation

The intent of the inclusion criteria was to be consistent with the superDimension Indications for Use.

| <u> </u> | · | · | · | · |
|----------|---|---|---|---|

The CIP will not be updated as the study has been closed by the sponsor and the Site IRBs.

| Name: Katie Bayliss | Role: Clinical Study Manager |
|-------------------------|---------------------------------------------|
| Signature: Katic Baylis | Date: $ 2 0 N 0 V 2 0 1 9 $ (dd/mmm/yyyy) |

Approved by:

| Name: Melody LaBeau | Role: Director of Clinical Affairs |
|---|---|
| Signature: WWW MWW | $Date: \underline{\mathcal{L}} \underline{\mathcal{O}} \underline{\mathcal{N}} \underline{\mathcal{O}} \underline{\mathcal{V}} \underline{\mathcal{L}} \underline{\mathcal{O}} \underline{\mathcal{I}} \underline{\mathcal{G}} (dd/mmm/yyyy)$ |